CLINICAL TRIAL: NCT02020603
Title: Efficacy of Hemostasis by Soft Coagulation Using Endoscopic Hemostatic Forceps in Comparison With Argon Plasma Coagulation for Acute Peptic Ulcer Bleeding
Brief Title: Efficacy of Hemostasis by Soft Coagulation Using Endoscopic Hemostatic Forceps for Acute Peptic Ulcer Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Wook Kim, Clinical fellow, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUB2013
Record Dates: First submitted 2013-12-15; First posted 2013-12-25 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Active Peptic Ulcer Disease/GI Bleeding
Keywords: peptic ulcer bleeding; hemostatic forceps; soft coagulation; argon plasma coagulation
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — Argon Plasma Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- APC group (Active Comparator): epinephrine injection plus argon plasma coagulation
  Interventions: Device: epinephrine injection plus argon plasma coagulation
- Forceps group (Active Comparator): epinephrine injection plus soft coagulation using hemostatic forceps
  Interventions: Device: epinephrine injection plus soft coagulation using hemostatic forceps

INTERVENTIONS:
Device: epinephrine injection plus soft coagulation using hemostatic forceps
  Arms: Forceps group
Device: epinephrine injection plus argon plasma coagulation
  Arms: APC group

SUMMARY:
Endoscopic high-frequency soft coagulation is available for the management of bleeding or nonbleeding visible vessels during endoscopic submucosal dissection. However, its efficacy on peptic ulcer bleeding has not been elucidated so far. The aim of this study was to evaluate the efficacy of hemostasis with soft coagulation using hemostatic forceps by comparing it with argon plasma coagulation (APC) in a prospective, randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* peptic ulcer with stigmata of recent hemorrhage

Exclusion Criteria:

* malignant ulcer
* previous gastric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Recurrence of bleeding within four weeks after initial hemostasis | up to 24 months

SECONDARY OUTCOMES:
initial hemostasis rate | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jae Young Jang, M.D., Study Chair — Kyung Hee University Hospital
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim JW, Jang JY, Lee CK, Shim JJ, Chang YW. Comparison of hemostatic forceps with soft coagulation versus argon plasma coagulation for bleeding peptic ulcer--a randomized trial. Endoscopy. 2015 Aug;47(8):680-7. doi: 10.1055/s-0034-1391565. Epub 2015 Mar 2. PMID 25730283